CLINICAL TRIAL: NCT07104084
Title: Comparison of Wound Healing Complications After Anterior Total Hip Arthroplasty Using Povidone-iodine or Chlorhexidine as Antiseptic Wash
Brief Title: Influence of Antiseptic Washes on Wound Healing Complications After THA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: F. Johannes Plate (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Sponsor-Investigator, F. Johannes Plate, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY25020138
Record Dates: First submitted 2025-07-27; First posted 2025-08-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hip Osteoarthritis; Avascular Necrosis of Femur Head
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Chlorhexidine washing solution (Experimental): Following component implantation a 3-minute chlorhexidine lavage followed by saline lavage will be performed.
  Interventions: Device: lavage chlorhexidine
- Povidone-iodine washing solution (Experimental): Following component implantation a 3-minute povidone-iodine lavage followed by saline lavage will be performed.
  Interventions: Device: lavage povidone-iodine

INTERVENTIONS:
Device: lavage chlorhexidine — Patient will receive a chlorhexidine lavage for 3 minutes following total hip component placement followed by saline lavage.
  Arms: Chlorhexidine washing solution
Device: lavage povidone-iodine — Patient will receive povidone-iodine lavage for 3 minutes following total hip component placement followed by saline lavage.
  Arms: Povidone-iodine washing solution

SUMMARY:
The purpose of this research trial is to evaluate the effect of two types of washing solutions on wound healing after total hip replacement surgery. Washing solutions are used routinely during total hip replacements to clean the wound after the components have been placed and the wound is about to be closed with sutures. It is currently not known which washing solution may be better for wound healing and whether a certain solution decreases the risk of wound healing complications after total hip replacement. Therefore, this research trial is being conducted.

Study participants will be randomized into one of two groups: washing the surgical wound with povidone-iodine solution (Surgiphor, Becton Dickinson, Franklin Lakes, NJ) or chlorhexidine solution (Irrisept, Irrimax Corporation, Lawrenceville, GA). All patients will undergo standard of care total hip replacements without any other change in surgery. The best type of solution that cleans the wound and potentially leads to better wound healing is unknown. This study will evaluate whether there is difference in surgical wound healing between the two washing solutions. The study will pay for the washing solutions. Patients will follow up for standard postoperative visits. At the 2-week and 6-week visits, pictures of the surgical incision will be taken and saved in the electronic medical record and evaluated in a standardized way for healing of the incision and the appearance of the scar. Postoperative complications and returns to the hospital or additional surgeries will be collected from the electronic medical record.

DETAILED DESCRIPTION:
Study participants will be randomized into one of two groups: washing the surgical wound with povidone-iodine solution (Surgiphor, Becton Dickinson, Franklin Lakes, NJ) or chlorhexidine solution (Irrisept, Irrimax Corporation, Lawrenceville, GA). All patients will undergo standard of care total hip replacements without any other change in surgery. The best type of solution that cleans the wound and potentially leads to better wound healing is unknown. This study will evaluate whether there is difference in surgical wound healing between the two washing solutions. Patients will follow up for standard postoperative visits. At the 2-week and 6-week visits, pictures of the surgical incision will be taken and saved in the electronic medical record and evaluated in a standardized way for healing of the incision and the appearance of the scar. Postoperative complications and returns to the hospital or additional surgeries will be collected from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis or avascular necrosis of the femoral head, failed conservative management, indicated for total hip replacement

Exclusion Criteria:

* reported or documented allergy to chlorhexidine or povidone-iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale | 2 weeks and 6 weeks postop
  The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability and surface area). All items are scored on a scale ranging from 1 ('like normal skin') to 10 ('worst scar imaginable'). The sum of the six items results in a total score of the POSAS observer scale. Categories boxes are added for each item. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location

SECONDARY OUTCOMES:
wound healing complications | up to 90 days from surgery
  drainage, dehiscence, suture abscess
Revision | up to 90 days from surgery
  Revision surgery, readmission

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Plate, MD, PhD, Principal Investigator — University of Pittsburgh; Frank J Plate, MD, PhD, Study Director — University of Pittsburgh; Frank J Plate, MD, PhD, Study Chair — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC East, Monroeville, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Anonymous outcomes comparing wound healing complication rates, revision and readmission rates with mean anonymous demographic data will be published.